CLINICAL TRIAL: NCT07239102
Title: A Real-World Clinical Retrospective Study of Firmonertinib in the Treatment of EGFR(+) NSCLC Patients With Central Nervous System Metastasis
Brief Title: Firmonertinib in the Treatment of EGFR(+) NSCLC Patients With Central Nervous System Metastasis
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HX-B-2025058
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; Central Nervous System Metastasis; Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EGFR-mutated NSCLC with brain metastases
  Interventions: Drug: Firmonertinib
- EGFR-mutated NSCLC with leptomeningeal metastases
  Interventions: Drug: Firmonertinib

INTERVENTIONS:
Drug: Firmonertinib — Firmonertinib any dose, oral

SUMMARY:
This is a clinical retrospective study that will collect and analyze clinical data from all patients treated with fumeitinib mesylate in the Oncology Department of Tiantan Hospital between January 1, 2020 and May 31, 2025. The data collection will include general demographic characteristics (gender, age, family history, smoking history, etc.), clinicopathological features, NGS test reports, fumeitinib initiation time and dosage, concomitant medications, local treatments (surgery, radiotherapy, etc.), and baseline and follow-up imaging examinations related to efficacy and safety. The study will conduct: 1) clinical data analysis; and 2) exploration of resistance-related clinical characteristics and influencing factors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage IIIb-IVb NSCLC or postoperative recurrent NSCLC;
2. Positive EGFR test result, which can be determined by methods such as RT-PCR/FISH/IHC/NGS from hospital laboratories or testing institutions;
3. Patients aged ≥18 years;
4. Patients have clinically received Firmonertinib treatment, with recorded objective efficacy evaluation and adverse reactions;
5. Sign the Beijing Tiantan Hospital broad informed consent form.

Exclusion Criteria:

- Patients who cannot provide follow-up data for at least one cycle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received at least one treatment cycle of Firmonertinib are defined as the Full Analysis Set (FAS). Except for specially specified study endpoints (such as DOR which is evaluated only in the population achieving objective response), the primary endpoints, secondary endpoints, and safety endpoints of the study are evaluated in the FAS.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
iPFS | From first dose until the event of interest, assessed between January 1, 2020 and May 30, 2025
  According to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) and the Response Assessment in Neuro-Oncology (RANO) criteria, the intracranial progression-free survival (iPFS) of Firmonertinib in subjects with advanced non-small cell lung cancer (NSCLC) with central nervous system (CNS) metastases and EGFR mutation-positive status will be evaluated separately for different cohorts

SECONDARY OUTCOMES:
iDCR | Within the study period from January 1, 2020 and May 30, 2025
  For different cohorts, evaluate the intracranial objective response rate (iORR) and disease control rate (iDCR) of Firmonertinib in subjects with advanced non-small cell lung cancer (NSCLC) positive for EGFR mutations and presenting with central nervous system metastases
PFS | From first dose until the event of interest, assessed between January 1, 2020 and May 30, 2025
  According to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) the progression-free survival (iPFS) of Firmonertinib in subjects with advanced non-small cell lung cancer (NSCLC) with central nervous system (CNS) metastases and EGFR mutation-positive status will be evaluated separately for different cohorts
OS | From first dose until death, assessed between January 1, 2020 and May 30, 2025
  measured from the date of first-line treatment initiation to the date of documented death
DOR | Within the study period from January 1, 2020 and May 30, 2025
  defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1 criteria, assessed at the first radiologic evaluation following initiation of treatment
TTR | assessed during the study period from January 1, 2020 and May 30, 2025.
  Defined as the time from the initiation of treatment to the date of first documented objective response (CR or PR) according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Li Xiaoyan, Beijing, Beijing Municipality, China